CLINICAL TRIAL: NCT00557700
Title: Study to Investigate the Effect of Inhaled Tiotropium Bromide on Neurokinin-A Induced Bronchoconstriction in Patients With Mild-to-moderate Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Guy Joos, MD, PhD, University Ghent
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2007/378
Record Dates: First submitted 2007-11-12; First posted 2007-11-14 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-06

CONDITIONS: Asthma
Keywords: Mild to moderate asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Administration of placebo
  Interventions: Drug: Administration of placebo
- 1 (Experimental): Administration of inhaled tiotropium bromide
  Interventions: Drug: Administration of inhaled tiotropium bromide

INTERVENTIONS:
Drug: Administration of inhaled tiotropium bromide — Administration of inhaled tiotropium bromide
  Arms: 1
Drug: Administration of placebo — Administration of placebo
  Arms: 2

SUMMARY:
This trial compares the outcome of treatment of mild to moderate asthma: inhaled tiotropium bromide versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Male or female, at least 18 years old
* Documented medical history of asthma (diagnosis at least 6 months ago)
* Non-smoker or at least stopped for 1 year (in case smoked earlier: maximum of 10 pack-years)
* Able to conduct a technically acceptable spirometry, methacholine and neurokinin-A provocation test.
* At visit 1: PC20 methacholine ≤ 8 mg/ml AND ≤ 3.3x10-7 mol/ml for the neurokinin-A provocation test.
* At visit 1: forced expiratory value in one second >= 80% of the predicted value.
* Female subjects may not get pregnant and should be using adequate contraception.

Exclusion Criteria:

* Airway infection within 6 weeks prior to first study visit.
* Other respiratory diseases (eg COPD, lung cancer, etc.)
* Participating in another clinical trial.
* Clinically relevant systemic diseases, other than asthma.
* Clinically significant laboratory deviations.
* Alcohol or drug abuse.
* Female subjects who are lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
The mean change in the provocative concentration of neurokinin-A (NKA) causing a 20% fall in the forced expiratory volume in one second (PC20NKA), as a measure of indirect airway hyperresponsiveness | After 20 days

SECONDARY OUTCOMES:
The change in the one-second-value in the forced vital capacity | After 20 days
The mean change in PC20 of methacholine, as a measure of direct airway hyperresponsiveness | After 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Guy Joos, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - University Hospital Ghent, Ghent
  - CHU Sart Tilman ULG, Liège

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be